CLINICAL TRIAL: NCT02553642
Title: A Prospectively Designed Study to Assess the Relationship Between Tumor Mutation Burden and Predicted Neo-antigen Burden in Patients With Advanced Melanoma or Bladder Cancer Treated With Nivolumab or Nivolumab Plus Ipilimumab (CA209-260)
Brief Title: Relationship Between Tumor Mutation Burden and Predicted Neo-antigen Burden in Patients With Advanced Melanoma or Bladder Cancer Treated With Nivolumab or Nivolumab Plus Ipilimumab (CA209-260)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: UConn Health (Other); Bristol-Myers Squibb (Industry); Adaptive Biotechnologies (Industry); MedGenome (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-126
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Melanoma
Keywords: Tumor Mutation; Nivolumab; Nivolumab plus Ipilimumab; Predicted Neo-antigen Burden; 15-126
MeSH Terms: conditions — Urinary Bladder Neoplasms; Melanoma | interventions — Nivolumab; Ipilimumab

ARMS (2):
- Melanoma Cancer Patients (Experimental): All eligible patients with melanoma will receive ipilimumab at a dose of 3 mg/kg combined with nivolumab at a dose of 1 mg/kg. The ipilimumab and nivolumab will be dosed every 3 weeks for 4 doses. Thereafter, patients may be eligible to continue to receive nivolumab monotherapy at a dose of 240 mg administered every 2 weeks OR nivolumab at dose of 480mg every 4 weeks for up to 2 years.
  Interventions: Drug: Nivolumab plus Ipilimumab
- Bladder Cancer Patients (Experimental): All eligible patients with bladder cancer will receive nivolumab at a dose of 240 mg administered every 2 weeks for up to 2 years, if the patient is clinically benefitting, the PI and treating investigator may elect to continue treatment beyond 2 years. All eligible patients with bladder cancer will receive nivolumab at a dose of 240 mg administered every 2 weeks for up to 2 years, if the patient is clinically benefitting, the PI and treating investigator may elect to continue treatment beyond 2 years.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Monotherapy Treatment - Nivolumab 240 mg flat dose Dosed q 2 weeks
  OR
  - Nivolumab 480 mg flat dose Dosed q 4 weeks
  for up to 2 years from 1st dose of nivolumab or until loss of clinical benefit
  Arms: Bladder Cancer Patients
Drug: Nivolumab plus Ipilimumab — Combination Treatment
  * Ipilimumab 3 mg/kg
  * Nivolumab 1 mg/kg Dosed q 3 weeks x 4 doses
  Arms: Melanoma Cancer Patients

SUMMARY:
The purpose of this study is to investigate the characteristics of tumors in patients treated with nivolumab and to identify features that help to predict a good or bad response to this drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB approved written informed consent in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
3. Pathologically confirmed locally advanced or metastatic disease per the treating institution's standard of care of the following tumor types

   Subjects with histologically confirmed locally advanced/unresectable or metastatic melanoma who meet all of the following criteria:

   i. Subjects have received any number of prior lines of therapy or may be treatment naïve ii. If the subject has been treated with a prior line of therapy, they must have had disease progression or be refractory to treatment

   OR

   b. Subjects with histologically or cytologically confirmed locally advanced/unresectable or metastatic urothelial carcinoma (including mixed histologies of urothelial carcinoma with elements of other subtypes) of the renal pelvis, ureter, bladder or urethra (referred to broadly in this protocol as "bladder cancer") who meet the following criteria: i. Subjects must have disease progression or refractory disease after their prior line of therapy. Subjects must have had at least 1 platinum based chemotherapy regimen for the treatment of metastatic or locally advanced unresectable disease. Subjects may have received any number of prior lines of therapy OR

   ii. Subjects with disease recurrence within 1 year of a platinum based neoadjuvant or adjuvant therapy for bladder cancer.

   OR

   iii. The subject actively refuses chemotherapy for the treatment of metastatic or locally advanced disease considered as standard treatment for this disease stage (i.e. a patient who has relapsed >1 year after treatment with neoadjuvant or adjuvant chemotherapy), despite being informed by the investigator about the treatment options. The subject's refusal must be documented.
4. Subjects must have measurable disease by CT scans or MRI per RECIST 1.1 criteria. Radiographic tumor assessment must be performed within 28 days prior to first dose of study drug.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Age ≥ 18 years.
7. Subjects must consent to allow for the acquisition of tumor sample prior to starting treatment on study (in most cases patients will require a tumor biopsy). This biopsy site may be the only site of measurable disease if the site is > 2 cm. The biopsy site must, in the opinion of the investigator, be likely to yield acceptable tumor sample for core biopsies as described in Appendix 4. It is also acceptable if tumor sample is obtained by excision biopsy or during surgery (i.e. if procedure was previously planned), provided the tumor sample can be processed as described in Appendix 4. In the case that a patient had a tumor sample acquired prior to consenting to the study and this tumor sample is acceptable for processing as described in Appendix 4 (i.e. frozen sample stored) and the tumor sample was acquired within 60 days of starting treatment, this is acceptable and a new biopsy will not be required.
8. Willingness to adhere to the study visit schedule and prohibitions as specified in this protocol.
9. Expected survival of at least 4 months.
10. At the time of day 1 of the study, patients must have completed chemotherapy, targeted therapy, investigational therapy, other immunotherapy, radiation therapy or major surgery (requiring general anesthesia) at least 28 days before administration of the first dose of nivolumab. Patients undergoing minor surgical procedures and biopsies that do not require general anesthesia may begin receiving study therapy if sufficiently recovered as determined by the treating investigator. Patients may have received prior focal radiotherapy for palliation of an isolated site of disease, which must be completed at least 14 days prior to day 1 of the study.

    Palliative (limited-field) radiation therapy is permitted during treatment with study drug (s), if all of the following criteria are met:
    1. The lesion being considered for palliative radiation is not a target lesion
    2. Radiation treatment is administered 12 weeks or greater after their first dose of study drug.
11. All baseline laboratory requirements will be assessed and should be obtained within 14 days of the first dose of study drug. Screening laboratory values must meet the following criteria:

White blood cells (WBCs) ≥ 2000/μL

Neutrophils ≥ 1000/μL

Platelets ≥ 100 x 103/μL

Hemoglobin ≥ 9.0 g/dL

Serum creatinine ≤ 1.5 x ULN (or glomerular filtration rate ≥ 40mL/min)

Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert's syndrome who must have total bilirubin ≤ 3.0mg/dL)

AST and ALT ≤ 3 x ULN

Albumin ≥ 3.0 g/dL

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases. Subjects with treated brain metastases are eligible if they meet all of the following criteria:

   1. Must be at least 28 days since craniotomy and resection, stereotactic radiosurgery, or whole brain radiotherapy.
   2. Must have no evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to first dose of study drug administration.
   3. Must have no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy or interfere with the interpretation of study results.
3. Other prior malignancy active within the previous 2 years except for local or organ confined early stage cancer that has been definitively treated with curative intent or does not require treatment, does not require ongoing treatment, has no evidence of active disease and has a negligible risk of recurrence and is therefore unlikely to interfere with the endpoints of the study.
4. Subjects with active autoimmune disease, symptoms or conditions. Subjects with vitiligo, type I diabetes, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, asymptomatic laboratory evidence of autoimmune disease (e.g.: +ANA, +RF, antithyroglobulin antibodies), or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses are permitted in the absence of active autoimmune disease.
6. Subjects who have received prior therapy with any T cell co-stimulation or checkpoint pathways such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-CD137; or other medicines specifically targeting T cells are prohibited. Prior therapy with BCG is permitted. Prior IL-2 is permitted.
7. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (CTCAE version 4) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy and which are not expected to resolve and result in long lasting sequelae such as neuropathy after platinum-based therapy, are permitted to enroll.
8. Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBV sAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection.
9. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. History of allergy to study drug component or history of severe hypersensitivity reaction to any monoclonal antibody
11. Women who are breast feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) done within 14 days of first dosing and urine test within 72 hours of first dosing.
12. Women of childbearing potential *(WOCBP) not using a medically acceptable means of contraception throughout the study treatment and for at least 23 weeks following the last dose of study treatment (5 half-lives of study drug plus 30 days duration of ovulatory cycle).

    *WOCBP are defined as those who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post-menopausal is defined as: Amenorrhea ≥ 12 consecutive months without another cause, or For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
13. Male subjects who are unwilling to use contraception during the treatment and for at least 31 weeks after the last dose of study treatment (5 half-lives of study drug plus 90 days duration of sperm turnover).
14. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Funt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- [Derived] Teo MY, Seier K, Ostrovnaya I, Regazzi AM, Kania BE, Moran MM, Cipolla CK, Bluth MJ, Chaim J, Al-Ahmadie H, Snyder A, Carlo MI, Solit DB, Berger MF, Funt S, Wolchok JD, Iyer G, Bajorin DF, Callahan MK, Rosenberg JE. Alterations in DNA Damage Response and Repair Genes as Potential Marker of Clinical Benefit From PD-1/PD-L1 Blockade in Advanced Urothelial Cancers. J Clin Oncol. 2018 Jun 10;36(17):1685-1694. doi: 10.1200/JCO.2017.75.7740. Epub 2018 Feb 28. PMID 29489427
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Melanoma Cancer Patients: All eligible patients with melanoma will receive ipilimumab at a dose of 3 mg/kg combined with nivolumab at a dose of 1 mg/kg. The ipilimumab and nivolumab will be dosed every 3 weeks for 4 doses. Thereafter, patients may be eligible to continue to receive nivolumab monotherapy at a dose of 240 mg administered every 2 weeks OR nivolumab at dose of 480mg every 4 weeks for up to 2 years.
  Nivolumab plus Ipilimumab: Combination Treatment
  * Ipilimumab 3 mg/kg
  * Nivolumab 1 mg/kg Dosed q 3 weeks x 4 doses
- Bladder Cancer Patients: All eligible patients with bladder cancer will receive nivolumab at a dose of 240 mg administered every 2 weeks for up to 2 years, if the patient is clinically benefitting, the PI and treating investigator may elect to continue treatment beyond 2 years. All eligible patients with bladder cancer will receive nivolumab at a dose of 240 mg administered every 2 weeks for up to 2 years, if the patient is clinically benefitting, the PI and treating investigator may elect to continue treatment beyond 2 years.
  Nivolumab: Monotherapy Treatment - Nivolumab 240 mg flat dose Dosed q 2 weeks
  OR
  - Nivolumab 480 mg flat dose Dosed q 4 weeks
  for up to 2 years from 1st dose of nivolumab or until loss of clinical benefit
Period: Overall Study
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients
Started | 10 | 71
Completed | 10 | 65
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Additional cancer dx | 0 | 1
Not completed — Never started treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients | Total
Number analyzed (Participants) | 10 | 69 | 79
Age, Continuous [Mean (Full Range); unit: years] | 60 [34 to 80] | 68 [41 to 90] | 67 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 14 | 18
  Male | 6 | 55 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 0 | 10
  Unknown or Not Reported | 0 | 68 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 55 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 8 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 69 | 79

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response in Bladder Cancer Participants to Nivolumab Monotherapy
Description: Primary clinical endpoint was proportion of patients who achieve a confirmed objective response rate (per RECIST 1.1) to nivolumab monotherapy in bladder cancer patients progressing on initial nivolumab monotherapy. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From treatment start, up to 2 years from initial dose of nivolumab.
Population: Only Bladder Cancer Patients were evaluated
Measure: Number (95% Confidence Interval); unit: percentage of participants with PR/CR
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients
Number analyzed (Participants) | 0 | 69
percentage of participants with PR/CR |  | 23 [14 to 35]

2. Primary Outcome: Confirmed Objective Response for Bladder Cancer Patients to Ipilimumab and Nivolumab Combination Therapy in Patients Progressing on Initial Nivolumab Monotherapy
Description: Primary clinical endpoint was proportion of patients who achieve a confirmed objective response rate (per RECIST 1.1) to ipilimumab and nivolumab combination therapy in bladder cancer patients progressing on initial nivolumab monotherapy.
Time Frame: From treatment start, up to 2 years from initial dose of nivolumab.
Population: Only Bladder Cancer Participants were evaluated
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients
Number analyzed (Participants) | 0 | 69
Participants
  Partial response + Complete response to ipilimumab and nivolumab combination therapy | 0 | 16
  No Partial response + Complete response to ipilimumab and nivolumab combo therapy | 0 | 53

3. Secondary Outcome: Tumor Mutational Burden for Evaluable Bladder Cancer Participants
Description: Primary correlative objective was to obtain information on mutational load and obtain preliminary prospective data on whether this factor is predictive of response to immunotherapy. Receiver operator characteristic (ROC) curves with mutational load as a continuous measure was used to estimate the area under the curve (AUC) to assess the detectability of responders. This was applicable to Bladder cohort.
Time Frame: At baseline
Population: Evaluable bladder cancer patients were analyzed
Measure: Median (Full Range); unit: mut/Mb
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients
Number analyzed (Participants) | 0 | 63
mut/Mb
  Median Tumor Mutational Burden/TMB among evaluable bladder participants |  | 502 [50 to 2255]
  TMB Missense Only |  | 92 [4 to 530]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Melanoma Cancer Patients | Bladder Cancer Patients
All-Cause Mortality (participants affected / at risk) | 2/10 | 51/69
Serious Adverse Events (participants affected / at risk) | 10/10 | 69/69
Other Adverse Events (participants affected / at risk) | 10/10 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Cancer Patients (N=10) | Bladder Cancer Patients (N=69)
Diarrhea (Gastrointestinal disorders) | 4 | 9
Colitis (Gastrointestinal disorders) | 2 | 0
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Resp, thoracic & mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Death NOS (General disorders) | 0 | 12
Acute Kidney Injury (Renal and urinary disorders) | 0 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Fatigue (General disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 4
Bladder Infection (Infections and infestations) | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3
Increased Alt (Investigations) | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 2
Increased Ast (Investigations) | 0 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 1
Bladder Flank Spams Bladder Burning (Renal and urinary disorders) | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Colonic Perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 1
Fever (General disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections and Infestations Other Specify Cellulitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pelvic Infection (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal Pain (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Weight Loss (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Cancer Patients (N=10) | Bladder Cancer Patients (N=69)
fatigue (General disorders) | 10 | 38
rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 31
Diarrhea (Gastrointestinal disorders) | 10 | 36
pruritus (Skin and subcutaneous tissue disorders) | 7 | 24
nausea (Gastrointestinal disorders) | 10 | 20
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 15
arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 14
anorexia (Metabolism and nutrition disorders) | 3 | 16
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 13
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 13
edema limbs (General disorders) | 0 | 10
hypothyroidism (Endocrine disorders) | 4 | 9
increased alt (Investigations) | 10 | 10
dry mouth (Gastrointestinal disorders) | 2 | 10
increased ast (Investigations) | 5 | 7
abdominal pain (Gastrointestinal disorders) | 6 | 5
fever (General disorders) | 5 | 6
hot flashes/night sweats (Vascular disorders) | 0 | 5
mucositis oral (Gastrointestinal disorders) | 0 | 6
constipation (Gastrointestinal disorders) | 0 | 5
dysgeusia (Nervous system disorders) | 0 | 5
headache (Nervous system disorders) | 0 | 4
infusion related reaction (Injury, poisoning and procedural complications) | 1 | 4
pain (General disorders) | 0 | 5
peripheral sensory neuropathy (Nervous system disorders) | 0 | 4
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 7
vomiting (Gastrointestinal disorders) | 5 | 2
chills (General disorders) | 0 | 6
dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
adrenal insufficiency (Endocrine disorders) | 3 | 2
colitis (Gastrointestinal disorders) | 1 | 3
Weight loss (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT02553642/Prot_SAP_000.pdf